CLINICAL TRIAL: NCT03525470
Title: Autonomic Adaptation to Hydration and Brain Functioning
Brief Title: Autonomic Adaptations to Hydration and Brain Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, David Benton, Professor, Swansea University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DB-0123-Hydration
Record Dates: First submitted 2018-04-13; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Hydration
Keywords: Hydration; Brain functioning; Heart-rate variability
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Cross-over design where on one occasion subjects lost 0.5% body weight,and drank 300ml water and on another occasion nothing was consumed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water (Experimental): Subjects consumed water
  Interventions: Biological: Water
- No water (Experimental): Subjects did not consume water
  Interventions: Other: No drink

INTERVENTIONS:
Biological: Water — 150 mil of water was drunk on two occasions
  Arms: Water
Other: No drink — Although body weight lost no drink consumed
  Arms: No water

SUMMARY:
The influence of relatively small decreases in hydration status have been little studied. On two occasions subjects will be allowed to lose about 0,5% of their body weight and one occasion 300ml of water will be consumed. Functional MRI will be used to monitor brain functioning when performing a mental arithmetic task. Heart rate variability will be monitored and related to differences in brain functioning when water has and has not been drunk

DETAILED DESCRIPTION:
On two mornings twelve male participants will be exposed to a temperature of 30oC for four hours and either drink or not drink two 150ml glasses of water during that time. The subjects the participate in an fMRI protocol during which they complete a modified version of the Paced Auditory Serial Addition Test (PASAT): a challenging arithmetic task designed to elicit autonomic arousal.

Throughout the morning subjects will their heart rate variability (HRV) monitored. At periodic intervals subjects will rate their thirst and mood by visual analogue scales and at the end of the PASAT task they rate its difficulty. Changes in body temperature and fluid loss (perspiration and urine) and urine osmolality will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Self declared as healthy and not taking any medication

Exclusion Criteria:

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
BOLD signal | One hour in scanner (1300-1400 hours)
  Participants will be presented with an arithmetic task, modified for use in the scanner, similar to the Paced Auditory Serial Addition Task: a 'stressful' task that measures calculation ability and is known to elicit an autonomic response 35. Pairs of two digit numbers appeared on a screen in red and participants will be required to mentally add or subtract the numbers. After 2 seconds the screens will be removed and a second screen appeared containing a correct and an incorrect answer. Participants will be required to press either a left or right button to indicate which answer was correct ). The speed of presentation is designed to be just at the level that it is possible to perform the task although it required mental effort and was 'stressful'.This allows investigation of areas of the brain associated with working memory but also those associated with emotional arousal.
Heart-rate variability | Differences on two testing occasions (0900 and 1300 hours) will be related to BOLD
  Differences in inter-beat intervals derived from RS800 Polar heart rate monitor with a sampling rate of 1000Hz. Profile to be analysed using the Kubios software

SECONDARY OUTCOMES:
Ratings of ,mood and perceived effort | Rated baseline (0830 hours), 30 mins later, 280 minutes later
  Using visual analogue scales mood and perceived effort will be rated.
Change in body weight | Measured at baseline (0830 hours), after 290 minutes (before urinating) and 300 mintues (after urinating)
  Scales, sensitive to 5 grams, will be used to monitor changes in body weight
Osmolality | Baseline (0830 hours) and after 300 minutes
  Using an Osmomat 300 freezing point osmometer the osmolality of urine will be measured at the beginning and end of testing sessions